CLINICAL TRIAL: NCT06839755
Title: The Prognostic Value of Positive Stress Echocardiography and Its Relationship with Invasive Coronary Angiography: the AMPHIPOLIS Study
Brief Title: The Positive Prognostic Value of Stress Echocardiography - AMPHIPOLIS STUDY
Acronym: AMPHIPOLIS
Status: Recruiting | Type: Observational
Sponsor: Hellenic Society of Cardiology (Other)
Collaborators: University of Cyprus (Other)
Responsible Party: Principal Investigator, Nikolaos Kadoglou, Assistant Professor of Cardiology, Hellenic Society of Cardiology
Other Study IDs: 20240901
Record Dates: First submitted 2025-02-04; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
Keywords: stress echocardiography; myocardial ischemia; prognosis; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with stress echocardiography positive for ischemia: patients with unknown and known CAD will undergo stress echocardiography for screening or monitoring purposes respectively.
  Patients with findings indicating myocardial ischemia will be considered eligible

SUMMARY:
This is a prospective, multicenter, observational study of patients with recent stress echocardiography positive for myocardial ischemia. Up to now 25 echocardiography labs form Greece and Cyprus have declared their intention to participate. The investigators will enroll 390 patients with a positive stress echo, who will undergo invasive coronary angiogram and then will be followed up for at least 6 months. The objectives are the following:

1. To assess the prognostic value of positive stress echo by monitoring for cardiovascular death and major adverse cardiovascular events (MACE) during the follow-up.
2. To investigate the relationship of stress echo findings with invasive coronary angiography anatomical findings.
3. The association of cardiovascular risk profile of participants with stress echo and coronary angiography findings.

DETAILED DESCRIPTION:
The stress echo-Amphipolis trial (NCT…) is a prospective, multicenter, self-controlled, open-label trial to evaluate the positive prognostic value of stress echocardiography and its relationship with ICA in patients with established or suspected coronary artery disease (CAD). The study is organized by the Working Group of Echocardiography (WGE) and it is endorsed by the Hellenic Cardiology Society (HCS), which has undertaken the structure of a common web-based platform to connect all echo labs.

Recruitment: The stress echo-Amphipolis trial will consecutively enroll adults with a positive SE based on echocardiographic findings. Then eligible patients will be asked to participate in the study and all their clinical and demographic parameters will be recorded in a web-based platform. Participants will undergo ICA within 6 weeks, and the results will be added in the platform. It will be conducted at 25 echocardiography labs in Greece and Cyprus. An open invitation has been previously sent to high-volume centers performing annually a significant number of SE (>250) to participate.

Therapy: Decision of therapy, either revascularization or conservative, will be at the discretion of the cardiologist of each patient. Post-SE pharmaceutical therapy will be prescribed in all patients according to current international guidelines.

Follow-up: Then patients will be followed up for at least 12 months to collect structured data regarding MACE: cardiovascular death, acute coronary syndromes (ACSs), revascularization interventions (re-stenosis or new cases of myocardial ischemia), developing symptoms (angina relapse or new onset). The time interval between SE and MACE will be recorded. Within follow-up period, all patients will be contacted by phone or with on-site visit for at least once. Surveillance data will be retrieved from medical records and patients will be asked for new symptoms onset of symptoms relapse. The total duration of the study is expected to be 2 years.

Committees: Besides this, the study will be monitored by 2 independent scientific groups: 1) The organizing committee (OC) consisting of the members of the core of the WGE, which will be responsible for the conduction of the study, data collection and monitoring/guiding of centers. 2) The Adjudication Committee (AC) which is comprised of cardiologists with high experience in SE coming from Greece and other countries. Moreover, written report and digital images should be available to the AC. This committee will decide in ambiguous cases of clinical endpoints achievement or will provide an expert opinion when there is a mismatch between SE and ICA findings. A 5% of cases will be randomly selected for a blind cross check from the AC.

Primary objectives

It is structured to investigate the following primary objectives:

1. The clinical outcomes-related to CAD in the long-term follow-up and their association with true positive and false positive results of SE. Up to now only a few large studies have examined the long-term occurrence of MACE, while two studies examined the prognostic value of false positive results of SE.
2. The relationship between functional (SE) and anatomical (ICA) findings and which parameters affect this relationship. Keeping ICA as the gold standard method for diagnosis of significant CAD, we will comparatively evaluated those modalities. A great advantage of the proposed study is to obtain the detailed information regarding medical therapy, type of revascularization and location of target vessel of patients with a positive SE result. Only a few studies have attempted a head-to-head comparison of those two different modalities concluding that SE and ICA are not the appropriate comparators for myocardial ischemia . Presumably, other factors or co-morbidities may considerably influence the functional behavior of stenotic coronary arteries. This has confused to some extent the decision-making work-up of interventional and non-interventional therapy of patients with CAD.
3. The long-term prognostic value of impaired CFR in case of either obstructed LAD stenosis or coronary microvascular disease (CMVD).

Secondary objectives

Additionally, the investigators have set some secondary objectives, since the large database will be available for subgroup analysis:

1. Investigation of the influence of certain conditions on the prognostic value and the ability of SE to detect significant coronary artery stenosis, like atrial fibrillation, bundle branch block, past revascularization, implanted pacemaker, traditional cardiovascular risk factors, medications during test (β-blockers, nitrates etc).
2. The association of related symptoms during test with the echocardiographic and ICA results. The relation of symptoms appearance during test with the diagnosis of CAD is subject of debate.
3. The comparative evaluation of SE and FFR findings, when they are available. Due to financial reasons, the FFR measurements will be obtained only when they are available.
4. The contributory role of SE to coronary microvascular disease (CMVD) diagnosis. The latter will be based on 4 criteria: a) symptoms of myocardial ischemia, (2) absence of obstructive CAD, (3) objective findings of myocardial ischemia (echocardiography and/or ECG) and (4) indication of impaired CFR.
5. Comparative evaluation of DSE and ESE in relation to prognostic value and relationship to ICA.

Study population - selection criteria The target group are adults with recent SE positive for myocardial ischemia regardless of its extent, symptoms during the test or previous history of CAD, who are keen to be followed-up for at least 1 year. Before SE the referral reasons can be suspected myocardial ischemia or screening of asymptomatic individuals with or without history of CAD. Underlying rhythm will not be a selection criterion, which means that in addition to individuals with sinus rhythm, patients presenting during the test atrial arrhythmias (fibrillation or flutter), frequent ventricular or supraventricular extra-systoles, bundle brunch block (BBB), pacing rhythm will be still eligible.

ELIGIBILITY:
Inclusion Criteria:

Patients with recent stress echocardiography positive for any extent of myocardial ischemia

Exclusion Criteria:

1. HFrEF requiring viability study.
2. Any symptomatic valvular disease causing symptoms.
3. Established or suspected cardiomyopathy.
4. Concomitant chronic diseases reducing life expectancy (active cancer, severe liver impairment, auto-immune diseases etc).
5. Recent acute coronary syndrome the last week.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known or unknown coronary artery disease, regardless of symptoms undergoing stress echocardiography.
Sampling Method: Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
cardiovascular death | 12 months
  The number of patients died during follow-up period due to cardiovascular reasons (e.g. myocardial infarction, stroke)
Major cardiovascular events | 12 months
  Number of patients presented with any of the following during the follow-up: acute coronary syndromes, new revascularization, angina recurrence or new myocardial ischemia diagnosis, arteries restenosis in interventional coronary angiography

SECONDARY OUTCOMES:
anatomical findings in coronary angiography | 12 months
  The number of coronary arteries with at least moderate stenosis (>50%) and the precise degree of anatomical stenosis in each of them according to coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Kadoglou, Principal Investigator — University of Cyprus
Locations (1):
- Hellenic Society of Cardiology, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
IPD are not to be shared with other researchers

REFERENCES:
- [Background] Picano E, Pierard L, Peteiro J, Djordjevic-Dikic A, Sade LE, Cortigiani L, Van De Heyning CM, Celutkiene J, Gaibazzi N, Ciampi Q, Senior R, Neskovic AN, Henein M. The clinical use of stress echocardiography in chronic coronary syndromes and beyond coronary artery disease: a clinical consensus statement from the European Association of Cardiovascular Imaging of the ESC. Eur Heart J Cardiovasc Imaging. 2024 Jan 29;25(2):e65-e90. doi: 10.1093/ehjci/jead250. PMID 37798126
- [Background] Woodward W, Dockerill C, McCourt A, Upton R, O'Driscoll J, Balkhausen K, Chandrasekaran B, Firoozan S, Kardos A, Wong K, Woodward G, Sarwar R, Sabharwal N, Benedetto E, Spagou N, Sharma R, Augustine D, Tsiachristas A, Senior R, Leeson P; EVAREST Investigators; EVAREST Investigators; Boardman H, d'Arcy J, Abraheem A, Banypersad S, Boos C, Bulugahapitiya S, Butts J, Coles D, Easaw J, Hamdan H, Jamil-Copley S, Kanaganayagam G, Mwambingu T, Pantazis A, Papachristidis A, Rajani R, Rasheed MA, Razvi NA, Rekhraj S, Ripley DP, Rose K, Scheuermann-Freestone M, Schofield R, Sultan A. Real-world performance and accuracy of stress echocardiography: the EVAREST observational multi-centre study. Eur Heart J Cardiovasc Imaging. 2022 Apr 18;23(5):689-698. doi: 10.1093/ehjci/jeab092. PMID 34148078
- [Background] Kadoglou NPE, Papadopoulos CH, Papadopoulos KG, Karagiannis S, Karabinos I, Loizos S, Theodosis-Georgilas A, Aggeli K, Keramida K, Klettas D, Kounas S, Makavos G, Ninios I, Ntalas I, Ikonomidis I, Sahpekidis V, Stefanidis A, Zaglavara T, Athanasopoulos G, Karatasakis G, Kyrzopoulos S, Kouris N, Patrianakos A, Paraskevaidis I, Rallidis L, Savvatis K, Tsiapras D, Nihoyannopoulos P. Updated knowledge and practical implementations of stress echocardiography in ischemic and non-ischemic cardiac diseases: An expert consensus of the Working Group of Echocardiography of the Hellenic Society of Cardiology. Hellenic J Cardiol. 2022 Mar-Apr;64:30-57. doi: 10.1016/j.hjc.2021.07.006. Epub 2021 Jul 28. PMID 34329766
- [Background] Zhuravleva OA, Ryabova TR, Vrublevsky AV, Svyazova NN, Margolis NY, Boshchenko AA. Stress Echocardiography by the ABCDE Protocol ln the Assessment of Prognosis of Stable Coronary Heart Disease. Kardiologiia. 2024 Apr 30;64(4):22-30. doi: 10.18087/cardio.2024.4.n2572. English, Russian. PMID 38742512